CLINICAL TRIAL: NCT02241356
Title: The Effect of Bifocals in Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R0002308; 2013-23 (Other Grant/Funding Number: Uitzicht)
Record Dates: First submitted 2014-08-29; First posted 2014-09-16 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Visual Acuity at Near; Accuracy of Accommodation; Prevention of Strabismus; Task Readiness
Keywords: Down syndrome; visual functions; bifocals; children; visual acuity at near
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single vision glasses (Active Comparator): single vision glasses
  Interventions: Device: single vision glasses
- bifocals (Experimental): bifocal glasses
  Interventions: Device: bifocals

INTERVENTIONS:
Device: bifocals — bifocal glasses with an addition of 2.5 Dioptres
  Other Names: bifocal glasses; reading glasses
  Arms: bifocals
Device: single vision glasses — single vision glasses
  Arms: single vision glasses

SUMMARY:
Visual acuity at near improves in children with Down syndrome using bifocals

DETAILED DESCRIPTION:
The accommodation is consistently reduced in 50 to 100% of children with Down syndrome and does not improve with age.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Down syndrome (DS)
* Accommodation lag >0.5 Dioptres for children with DS <12 years and >0.75 Dioptres for children older than age 12 or Visual acuity at near is worse than at distance and >0.1
* Age range 2-14 years
* Speaks Dutch as the first language
* Must be verbal or able to understand instructions
* Must be able to perform a task sitting on a chair and working at a table

Exclusion Criteria:

* Visual acuity at near < 0.1
* Not able to do vision tests at age over 5
* Has worn bifocals already
* Other significant eye diseases, such as keratoconus, cataract or high myopia (>S-6.00).
* Diagnoses of any neurological, sensory or behavioural disorders such as autism, microcephaly or significant hearing loss.
* Prematurity, born premature after a pregnancy term less than 36 weeks
* Born after severe perinatal problems

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
• Change from baseline in visual acuity at near measured in decimals and in Logarithm of the Minimum Angle of Resolution (LogMAR) at 16 months. | baseline to 12 months later
  visual acuity is measured in decimals and in Logarithm of the Minimum Angle of Resolution (LogMAR) at baseline and at the end of the study 16 months later. We will calculate the difference.

SECONDARY OUTCOMES:
• Visual acuity at near measured in decimals and in Logarithm of the Minimum Angle of Resolution (LogMAR) at 16 months. | after 12 months
  visual acuity at near measured in decimals and in Logarithm of the Minimum Angle of Resolution (LogMAR) at 16 months.
• Change from baseline in visual acuity at distance measured in decimals and in Logarithm of the Minimum Angle of Resolution (LogMAR) at 16 months. | baseline to 12 months later
  Visual acuity at distance is measured in decimals and in Logarithm of the Minimum Angle of Resolution (LogMAR) at baseline and at the end of the study 16 months later. We will calculate the difference.
• Change from baseline in accuracy of accommodation response measured in Dioptres. | baseline to 12 months later
  We will measure the accuracy of accommodation in Dioptres at baseline and after 16 months. We will calculate the difference.
• Change in percentage of participants with strabismus | baseline to 12 months later
  We will calculate the percentage of participants with strabismus at baseline and at the end of the study, 16 months later. Then we can calculate the difference in percentage of participants with strabismus.
• Change in score of task readiness of the children | baseline to 12 months later
  We will measure task readiness in scores of attention, reaction time, inhibition and working memory at baseline and at the end of the study 16 months later. Then we calculate the difference in this score.

OTHER OUTCOMES:
• Possible prognostic determinants at baseline for improvement of visual acuity at near | participants will be followed for the duration of 12 months, after the last included participant has been followed up for 18 months we will do this analysis
  Applying a multivariate logistic regression model using a backward variable elimination procedure (selection criterion P < 0.05, removal criterion P < 0.10) to test a key set of independent prognostic variables (measured at baseline) for better visual acuity at near after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: H HL Goossens, PhD, Principal Investigator — Radboudumc, Dept. Cognitive Neuroscience/126
Locations (1):
- Isala Hospital, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Background] Nandakumar K, Leat SJ. Bifocals in children with Down syndrome (BiDS) - visual acuity, accommodation and early literacy skills. Acta Ophthalmol. 2010 Sep;88(6):e196-204. doi: 10.1111/j.1755-3768.2010.01944.x. PMID 20626718
- [Background] Al-Bagdady M, Stewart RE, Watts P, Murphy PJ, Woodhouse JM. Bifocals and Down's syndrome: correction or treatment? Ophthalmic Physiol Opt. 2009 Jul;29(4):416-21. doi: 10.1111/j.1475-1313.2009.00646.x. Epub 2009 May 11. PMID 19470088
- [Background] Cregg M, Woodhouse JM, Pakeman VH, Saunders KJ, Gunter HL, Parker M, Fraser WI, Sastry P. Accommodation and refractive error in children with Down syndrome: cross-sectional and longitudinal studies. Invest Ophthalmol Vis Sci. 2001 Jan;42(1):55-63. PMID 11133848